CLINICAL TRIAL: NCT04148833
Title: Treatment of Patients With Coronary and Aortic Atherosclerotic Disease With Paclitaxel-associated to LDL Like Nanoparticles. A Randomized, Double-blind, Placebo-control Trial.
Brief Title: Treatment of Patients With Atherosclerotic Disease With Paclitaxel-associated to LDL Like Nanoparticles
Acronym: PAC-MAN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Raul Cavalcante Maranhão, Head Professor of Clinical Biochemistry, Faculty of Pharmaceutical Sciences; Director, Lipid Metabolism Laboratory, Heart Institute of the Medical School, University of São Paulo, São Paulo, Brazil. MD, PHD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02090118.7.0000.0068
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Inflammation
Keywords: ATHEROSCLEROSIS; CORONARY ARTERY DISEASE; INFLAMATION; NANOPARTICLES; PACLITAXEL; DRUG TARGETING; DRUG DELIVERY SYSTEM
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDE-Paclitaxel (Experimental): Paclitaxel carried by a lipid nanoparticle (LDE-Paclitaxel)
  Interventions: Drug: LDE-Paclitaxel
- LDE-Placebo (Placebo Comparator): Lipid nanoparticle (LDE)
  Interventions: Drug: LDE-Placebo

INTERVENTIONS:
Drug: LDE-Paclitaxel — LDE-Paclitaxel at the dose of 175 mg/m2 IV each 21 days for 6 weeks
  Arms: LDE-Paclitaxel
Drug: LDE-Placebo — LDE-Placebo at the dose of 175 mg/m2 IV each 21 days for 6 weeks
  Arms: LDE-Placebo

SUMMARY:
The investigators propose a prospective, randomized, double-blind, placebo-controlled study. The purpose of the study is to evaluate the safety and efficacy of an anti-proliferative agent paclitaxel in a cholesterol-rich non-protein nanoparticle (Paclitaxel -LDE) in patients with stable coronary disease.

Patients with multi-vessels stable coronary disease will be randomized to receive Paclitaxel-LDE IV or placebo-LDE IV each 21 days for 6 weeks. The primary and main secondary endpoints will be analyzed by coronary and aortic CTA, that will be performed 1-4 weeks after randomization and at 3-8 weeks after the last treatment cycle.

Patients will undergo clinical and laboratory safety evaluations before each treatment cycle and 3-8 weeks after the last cycle. An algorithm for drug suspension based on clinical and laboratory finding will be followed.

DETAILED DESCRIPTION:
Atherosclerosis is a life-threatening condition, as long as cardiovascular disease is responsible for 31% of all global mortality.

Inflammation is extremely important in atherosclerosis pathophysiology. The use of inflammatory biomarkers to predict risk, monitor treatments and guide therapy, has shown substantial potential for clinical applicability. Many studies in primary and secondary prevention of cardiovascular disease showed that individuals with lower high sensitive C-reactive protein (hsCRP) have better clinical outcomes than those with higher levels. The potential benefit of anti-inflammatory therapy in atherosclerosis has been previously demonstrated in studies in patients with chronic inflammatory diseases, such as rheumatoid arthritis (AR); in systemic lupus erythematosus; in psoriasis and inflammatory bowel disease, in this patients the spread of the inflammatory cascade results in premature atherosclerotic plaque formation. Cardiovascular mortality is the cause of death in 40-50% of AR patients. The treatment of systemic diseases with TNF-a inhibitors has been associated with a reduction in cardiovascular events in patients with AR and psoriasis.

In this setting, the use of non-invasive treatments to reduce lesion size and inflammation is essential for the prevention of sub-sequent cardiovascular events.

The most potent anti-proliferative drugs currently available are chemotherapeutic agents used for cancer treatment. However, the systemic use of these drugs at high doses for the treatment of atherosclerotic cardiovascular diseases is unlikely due to their significant, often life-threatening toxicity. Nonetheless, the toxicity of such agents can be strongly diminished by the use of optimized drug-delivery systems. In a pioneer study performed on patients with acute leukemia, Maranhão et al. reported the potential of a cholesterol-rich non-protein nanoparticle (LDE) as a drug targeting agent. LDE particles have lipid compositions and structures that resemble low-density lipoprotein (LDL) and can be injected directly into the bloodstream. When LDE particles come into contact with plasma, the particles acquire exchangeable apolipoproteins from native lipoproteins, such as apolipoprotein (apo) E, which binds the particles to LDL receptors. In neoplastic cells, lipoprotein receptors are overexpressed, such that uptake of native LDL and of LDE particles is increased relative to that in normal tissues. In aortas of cholesterol-fed rabbits the uptake of LDE particles is increased in comparison to normal aortas and in rabbit-grafted hearts take up the nanoemulsion at amounts fourfold greater than native hearts.

LDE-paclitaxel treatment of rabbits induced to exhibit atherosclerosis via high cholesterol intake resulted in a 65% reduction in lesion size. In rabbits that underwent heterotopic heart transplantation, LDE-paclitaxel treatment markedly reduced heart graft damage by preventing coronary vessel destruction and macrophage invasion into the myocardium.

In a pilot study Maranhão et al showed that treatment with high-dose LDE-paclitaxel had low enough toxicity to permits the use in patients with cardiovascular disease, and an average 18% reduction in aortic plaque volume in four out of the eight participants, which is a promising finding. This result was especially noteworthy in view of the short 18-week treatment period and when considering that plaque reduction did not occur in any of the control group patients. In contrast, statistically significant disease progression was observed in the non-treated control patients.

The aim of this study is to investigate whether patients with aortic and coronary atherosclerotic disease showed good tolerability to LDE-paclitaxel treatment and whether this formulation could achieve reduction in plaque volume and characteristics by coronary and aortic CT angiography.

ELIGIBILITY:
Inclusion Criteria:

* Multi-vessels coronary artery disease diagnosis by coronary CTA scan or invasive angiography
* Aortic atherosclerosis diagnosis by multidetector computed tomography (MDCT) angiography.
* Signing the study informed consent.

Exclusion Criteria:

* History of AMI in the last 30 days
* Heart failure with ejection fraction <40%
* Estimated glomerular filtration rate < 40 mL/min/1.73 m2.
* Prior history of chronic infectious disease, including tuberculosis, severe fungal disease, or known HIV positive.
* Chronic hepatitis B or C infection.
* Prior history of nonbasal cell malignancy or myeloproliferative or lymphoproliferative disease within the past 5 years.
* White blood cell count <4000/mm3, hematocrit <32%, or platelet count <75000/mm3.
* Alanine aminotransferase levels (ALT) greater than 3-fold the upper limit of normal.
* History of actual alcohol abuse or unwillingness to limit alcohol consumption to < 4 drinks per week.
* Pregnancy or breastfeeding.
* Women of child bearing potential, even if currently using contraception.
* Men who plan to father children during the study period or who are unwilling to use contraception.
* Chronic use of oral steroid therapy or other immunosuppressive or biologic response modifiers.
* Known chronic pericardial effusion, pleural effusion, or ascites.
* Angina pectoris CCS III-IV
* New York Heart Association class III-IV congestive heart failure.
* Contraindication for the use of iodinated contrast
* Life expectancy of < 1 years.
* Acute or Chronic aortic dissection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-23 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2021-08-23 (Estimated)

PRIMARY OUTCOMES:
Low Attenuation Plaque Volume (LAPV) coronary | Baseline and change from baseline to 6-8 months
  Compare Low attenuation Plaque Volume( LAPV) measured by coronary CTA between Paclitaxel-LDE and Placebo-LDE groups.
Low Attenuation Plaque Volume (LAPV) aortic | Baseline and change from baseline to 6-8 months
  Compare Low attenuation Plaque Volume( LAPV) measured by aortic CTA between Paclitaxel-LDE and Placebo-LDE groups.

SECONDARY OUTCOMES:
Noncalcified plaque volume (NCPV) | Baseline and change from baseline to 6-8 months
  Compare Noncalcified plaque volume (NCPV) measured by coronary CTA between Paclitaxel-LDE and Placebo-LDE groups.
Dense calcified plaque volume (DCPV) | Baseline and change from baseline to 6-8 months
  Compare Dense calcified plaque volume (DCPV) measured by coronary CTA between Paclitaxel-LDE and Placebo-LDE groups.
Total lumen value (TLV) | Baseline and change from baseline to 6-8 months
  Compare Total lumen value (TLV) measured by coronary CTA between Paclitaxel-LDE and Placebo-LDE groups.
Remodeling index (RI) | Baseline and change from baseline to 6-8 months
  Compare Remodeling index (RI)measured by coronary CTA between Paclitaxel-LDE and Placebo-LDE groups.
Perivascular fat attenuation index (FAI) | Baseline and change from baseline to 6-8 months
  Compare Perivascular fat attenuation index (FAI)measured by coronary CTA between Paclitaxel-LDE and Placebo-LDE groups.
Total atheroma volume (TAV) | Baseline and change from baseline to 6-8 months
  Compare Total atheroma volume (TAV) measured by coronary CTA between Paclitaxel-LDE and Placebo-LDE groups.
Total atheroma volume (TAV) aortic | Baseline and change from baseline to 6-8 months
  Compare Total atheroma volume (TAV) measured by aortic CTA between Paclitaxel-LDE and Placebo-LDE groups.
Clinical significant symptoms | 3±1, 6±1, 9±1, 12±1, 15±1 and 18±1 weeks
  Compare the incidence of clinical significant symptoms (new and persistent stomatitis, vomiting, diarrhea, unexplained cough with fever, shortness of breath, alopecia, neurotoxicity, myalgia, arthralgias, bradycardia, hypotension, local pain) reported in each visit between Paclitaxel-LDE and Placebo-LDE groups.
Other adverse events | 3±1, 6±1, 9±1, 12±1, 15±1 and 18±1 weeks
  Compare the incidence of other adverse events (not expected) reported in each visit between Paclitaxel-LDE and Placebo-LDE groups.
Red blood cell count | 3±1, 6±1, 9±1, 12±1, 15±1 and 18±1 weeks
  Compare hemoglobin and hematocrits levels between Paclitaxel-LDE and Placebo-LDE groups.
White blood cell count | 3±1, 6±1, 9±1, 12±1, 15±1 and 18±1 weeks
  Compare leucocyte and neutrophil levels levels between Paclitaxel-LDE and Placebo-LDE groups.
Platelet count | 3±1, 6±1, 9±1, 12±1, 15±1 and 18±1 weeks
  Compare total Platelet levels between Paclitaxel-LDE and Placebo-LDE groups.
Alanine aminotransferase (ALT) | 3±1, 6±1, 9±1, 12±1, 15±1 and 18±1 weeks
  Compare Alanine aminotransferase (ALT) levels between Paclitaxel-LDE and Placebo-LDE groups.
Aspartate aminotransferase (AST) | 3±1, 6±1, 9±1, 12±1, 15±1 and 18±1 weeks
  Compare Aspartate aminotransferase (AST) levels between Paclitaxel-LDE and Placebo-LDE groups.
Creatinine | 3±1, 6±1, 9±1, 12±1, 15±1 and 18±1 weeks
  Compare Creatinine levels between Paclitaxel-LDE and Placebo-LDE groups.
Urea | 3±1, 6±1, 9±1, 12±1, 15±1 and 18±1 weeks
  Compare Urea levels between Paclitaxel-LDE and Placebo-LDE groups.

OTHER OUTCOMES:
High-sensitivity C reactive protein (hs-CRP) | Baseline and change from baseline to 6-8 months
  Compare High-sensitivity C reactive protein (hs-CRP) between Paclitaxel-LDE and Placebo-LDE groups.
Interleukin 6 (IL-6) | Baseline and change from baseline to 6-8 months
  Compare Interleukin 6 (IL-6) between Paclitaxel-LDE and Placebo-LDE groups.
Interleukin 1b (IL-1b) | Baseline and change from baseline to 6-8 months
  Compare Interleukin 1b (IL-1b) between Paclitaxel-LDE and Placebo-LDE groups.
Interleukin 10 (IL-10) | Baseline and change from baseline to 6-8 months
  Compare Interleukin 10 (IL-10) between Paclitaxel-LDE and Placebo-LDE groups.
Interleukin 8 (IL-8) | Baseline and change from baseline to 6-8 months
  Compare Interleukin 8 (IL-8) between Paclitaxel-LDE and Placebo-LDE groups.
Interferon gamma (IFN-y) | Baseline and change from baseline to 6-8 months
  Compare Interferon gamma (IFN-y) between Paclitaxel-LDE and Placebo-LDE groups.
Tumor necrosis factor-alpha (TNF-a) | Baseline and change from baseline to 6-8 months
  Compare Tumor necrosis factor-alpha (TNF-a) between Paclitaxel-LDE and Placebo-LDE groups.
Total Cholesterol | Baseline and change from baseline to 6-8 months
  Compare Total Cholesterol levels between Paclitaxel-LDE and Placebo-LDE groups.
High-density lipoprotein cholesterol (HDL) | Baseline and change from baseline to 6-8 months
  Compare High-density lipoprotein cholesterol (HDL) levels between Paclitaxel-LDE and Placebo-LDE groups.
Low-density lipoprotein cholesterol (LDL) | Baseline and change from baseline to 6-8 months
  Compare Low-density lipoprotein cholesterol (LDL) levels between Paclitaxel-LDE and Placebo-LDE groups.
Triglyceride | Baseline and change from baseline to 6-8 months
  Compare Triglyceride levels between Paclitaxel-LDE and Placebo-LDE groups.
Creatine phosphokinase (CPK) | Baseline and change from baseline to 6-8 months
  Compare Creatine phosphokinase (CPK) levels between Paclitaxel-LDE and Placebo-LDE groups.
Cholesterol efflux | Baseline and change from baseline to 6-8 months
  Compare Cholesterol efflux between Paclitaxel-LDE and Placebo-LDE groups.

CONTACTS AND LOCATIONS:
Overall Officials: Raul C Maranhão, MD;PhD, Study Chair — Director Lipid Metabolism Laboratory, Heart Institute
Locations (1):
- Heart Institute (InCor) - University of São Paulo Medical School, São Paulo, Brazil, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shapiro MD, Fazio S. From Lipids to Inflammation: New Approaches to Reducing Atherosclerotic Risk. Circ Res. 2016 Feb 19;118(4):732-49. doi: 10.1161/CIRCRESAHA.115.306471. PMID 26892970
- [Background] van Diepen JA, Berbee JF, Havekes LM, Rensen PC. Interactions between inflammation and lipid metabolism: relevance for efficacy of anti-inflammatory drugs in the treatment of atherosclerosis. Atherosclerosis. 2013 Jun;228(2):306-15. doi: 10.1016/j.atherosclerosis.2013.02.028. Epub 2013 Mar 1. PMID 23518178
- [Background] Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Study Group. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med. 2008 Nov 20;359(21):2195-207. doi: 10.1056/NEJMoa0807646. Epub 2008 Nov 9. PMID 18997196
- [Background] Ridker PM. Residual inflammatory risk: addressing the obverse side of the atherosclerosis prevention coin. Eur Heart J. 2016 Jun 7;37(22):1720-2. doi: 10.1093/eurheartj/ehw024. Epub 2016 Feb 22. No abstract available. PMID 26908943
- [Background] Khan R, Spagnoli V, Tardif JC, L'Allier PL. Novel anti-inflammatory therapies for the treatment of atherosclerosis. Atherosclerosis. 2015 Jun;240(2):497-509. doi: 10.1016/j.atherosclerosis.2015.04.783. Epub 2015 Apr 18. PMID 25917947
- [Background] Prodanovich S, Ma F, Taylor JR, Pezon C, Fasihi T, Kirsner RS. Methotrexate reduces incidence of vascular diseases in veterans with psoriasis or rheumatoid arthritis. J Am Acad Dermatol. 2005 Feb;52(2):262-7. doi: 10.1016/j.jaad.2004.06.017. PMID 15692471
- [Background] Barnabe C, Martin BJ, Ghali WA. Systematic review and meta-analysis: anti-tumor necrosis factor alpha therapy and cardiovascular events in rheumatoid arthritis. Arthritis Care Res (Hoboken). 2011 Apr;63(4):522-9. doi: 10.1002/acr.20371. PMID 20957658
- [Background] Vaidya K, Arnott C, Martinez GJ, Ng B, McCormack S, Sullivan DR, Celermajer DS, Patel S. Colchicine Therapy and Plaque Stabilization in Patients With Acute Coronary Syndrome: A CT Coronary Angiography Study. JACC Cardiovasc Imaging. 2018 Feb;11(2 Pt 2):305-316. doi: 10.1016/j.jcmg.2017.08.013. Epub 2017 Oct 18. PMID 29055633
- [Background] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Background] Dias ML, Carvalho JP, Rodrigues DG, Graziani SR, Maranhao RC. Pharmacokinetics and tumor uptake of a derivatized form of paclitaxel associated to a cholesterol-rich nanoemulsion (LDE) in patients with gynecologic cancers. Cancer Chemother Pharmacol. 2007 Jan;59(1):105-11. doi: 10.1007/s00280-006-0252-3. Epub 2006 May 13. PMID 16699792
- [Result] Solomon DH, Karlson EW, Rimm EB, Cannuscio CC, Mandl LA, Manson JE, Stampfer MJ, Curhan GC. Cardiovascular morbidity and mortality in women diagnosed with rheumatoid arthritis. Circulation. 2003 Mar 11;107(9):1303-7. doi: 10.1161/01.cir.0000054612.26458.b2. PMID 12628952
- [Result] Maranhao RC, Vital CG, Tavoni TM, Graziani SR. Clinical experience with drug delivery systems as tools to decrease the toxicity of anticancer chemotherapeutic agents. Expert Opin Drug Deliv. 2017 Oct;14(10):1217-1226. doi: 10.1080/17425247.2017.1276560. Epub 2017 Jan 1. PMID 28042707
- [Result] Maranhao RC, Tavares ER, Padoveze AF, Valduga CJ, Rodrigues DG, Pereira MD. Paclitaxel associated with cholesterol-rich nanoemulsions promotes atherosclerosis regression in the rabbit. Atherosclerosis. 2008 Apr;197(2):959-66. doi: 10.1016/j.atherosclerosis.2007.12.051. Epub 2008 Mar 4. PMID 18289548
- [Result] Shiozaki AA, Senra T, Morikawa AT, Deus DF, Paladino-Filho AT, Pinto IM, Maranhao RC. Treatment of patients with aortic atherosclerotic disease with paclitaxel-associated lipid nanoparticles. Clinics (Sao Paulo). 2016 Aug;71(8):435-9. doi: 10.6061/clinics/2016(08)05. PMID 27626473
- [Result] Maranhao RC, Garicochea B, Silva EL, Llacer PD, Pileggi FJ, Chamone DA. Increased plasma removal of microemulsions resembling the lipid phase of low-density lipoproteins (LDL) in patients with acute myeloid leukemia: a possible new strategy for the treatment of the disease. Braz J Med Biol Res. 1992;25(10):1003-7. PMID 1342820
- [Result] Lourenco-Filho DD, Maranhao RC, Mendez-Contreras CA, Tavares ER, Freitas FR, Stolf NA. An artificial nanoemulsion carrying paclitaxel decreases the transplant heart vascular disease: a study in a rabbit graft model. J Thorac Cardiovasc Surg. 2011 Jun;141(6):1522-8. doi: 10.1016/j.jtcvs.2010.08.032. Epub 2011 Mar 31. PMID 21458008
- [Derived] Marinho LL, Rached FH, Morikawa AT, Tavoni TM, Cardoso APT, Torres RVA, Assuncao AN Jr, Serrano CV Jr, Nomura CH, Maranhao RC. Safety and possible anti-inflammatory effect of paclitaxel associated with LDL-like nanoparticles (LDE) in patients with chronic coronary artery disease: a double-blind, placebo-controlled pilot study. Front Cardiovasc Med. 2024 Feb 21;11:1342832. doi: 10.3389/fcvm.2024.1342832. eCollection 2024. PMID 38450375
- See also: WHO — http://www.who.int/mediacentre/factsheets/fs317/en/